CLINICAL TRIAL: NCT05488639
Title: Injury and Illness Surveillance at FIFA U-17 & U-20 Women's World Cups.
Status: Suspended | Type: Observational
Why Stopped: Insufficient participation
Sponsor: Federation Internationale de Football Association (Other)
Responsible Party: Sponsor
Other Study IDs: 1
Record Dates: First submitted 2022-08-03; First posted 2022-08-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Injuries; Illness
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Football players at the FIFA U-20 Women's World Cup 2022.: * Upper age limit: all players must be a maximum of 20 years old by the end of the calendar year in which the World Cup 2022 is played (i.e. all players of the teams were born on or after 1 January 2002).
  * Lower age limit: all players must be at least 16 years old by the end of the calendar year in which the World Cup 2022 is played (i.e. all players of the teams were born on or before 31 December 2006).
  Interventions: Other: Registration of football exposure and occurrence of injuries and illnesses only
- Football players at the FIFA U-17 Women's World Cup 2022.: * Upper age limit: all players must be a maximum of 17 years old by the end of the calendar year in which the World Cup 2022 is played (i.e. all players of the teams were born on or after 1 January 2005).
  * Lower age limit: all players must be at least 15 years old by the end of the calendar year in which the World Cup 2022 is played (i.e. all players of the teams were born on or before 31 December 2007).
  Interventions: Other: Registration of football exposure and occurrence of injuries and illnesses only

INTERVENTIONS:
Other: Registration of football exposure and occurrence of injuries and illnesses only — Injury & illness registration
  Data on injury and illness is gathered following the recommended methodology in the football extension of the International Olympic Committee consensus statement on methods for recording and reporting of epidemiological data on injury and illness in sport. This includes characteristics such as mode of onset, injury mechanism, diagnosis and classification according to body area, tissue, and pathology type, and illness categories for organ system and etiology. Time-loss will be counted in number of days.

SUMMARY:
The primary objective is to provide an overview of the incidence and characteristics of time-loss injuries and illnesses during the FIFA U-20 and U-17 Women's World Cups in 2022.

DETAILED DESCRIPTION:
This research project will be performed at the FIFA U-20 Women's World Cup 2022 final tournament which is played in Alajuela and San José, Costa Rica between August 10 and August 28, 2022, and the FIFA U-17 Women's World Cup 2022 final tournament which is played in Bhubaneswar, Goa, and Navi Mumbai, India between October 11 and October 30th, 2022.

Each tournament includes 16 national teams, and each team is allowed to select 21 players, giving at total of 336 potential participants per tournament. In total, 32 matches will be played over 19 days, with the 24 group stage matches played in the first 8 days and the 8 knock-out matches played in the last 9 days.

Study duration The study will start from the first day of training with the national team prior the tournament until the day of the last match of the tournament. Consequently, the number of recordings will vary between teams depending on the duration of their pre-tournament training (usually 1-3 weeks), and their performance and progression through the tournament. In order to assess the severity of injuries (based on the length of time a player is unable to play for), all injuries are to be recorded until they are fully rehabilitated, even if this is after the end of the tournament. Each contact person therefore also needs to report when an injured player who has left the tournament has returned to full training with their club team after the tournament.

Demographic information Individual demographic information, including age, height, weight, playing position, and leg dominance (preferred kicking leg), is collected following inclusion.

Injury & illness registration Data on injury and illness is gathered following the recommended methodology in the football extension of the International Olympic Committee consensus statement on methods for recording and reporting of epidemiological data on injury and illness in sport.10 This includes characteristics such as mode of onset, injury mechanism, diagnosis and classification according to body area, tissue, and pathology type, and illness categories for organ system and etiology. Time-loss will be counted in number of days.

Exposure registration Training and match exposure will be recorded in minutes for each participant on a weekly basis for the duration of the tournament. Training exposure includes for example any sports-specific training, strength and conditioning sessions, and active recovery sessions. Illness exposure will be recorded in days for each participant from their first day of training until their last match.

The primary objective is to provide an overview of the incidence and characteristics of time-loss injuries and illnesses during the FIFA U-20 and U-17 Women's World Cups in 2022.

A secondary objective is to explore any differences in injury characteristics between the two age categories.

The primary variables of interest are time-loss injuries and time-loss illnesses.

* Time-loss is defined as inability of a player to complete the current or future training session or match.
* Injury is defined as tissue damage or other derangement of normal physical function resulting from rapid or repetitive transfer of kinetic energy.
* Illness is defined as a health-related complaint or disorder experienced by an athlete, not considered as an injury.

Descriptive statistics is used to provide an overview of the participant demographics and injury and illness occurrence. Injury incidence is calculated as number of injuries per 1000 hours of exposure, and injury burden is calculated as time-loss days per 1000 hours of exposure. Injury incidence and burden will be reported for training and match injuries separately. Illness incidence is calculated per 365 exposure days. Potential age group comparison in burden will be performed using an independent t-test/Mann-Whitney U Test depending on data distribution. Potential missing data will be excluded from analysis and reported accordingly.

Sample size No a priori sample size calculation is performed as we will attempt to include all eligible participants from the two tournaments giving a total possible sample size of 672 female football players.

ELIGIBILITY:
Inclusion Criteria:

* All participating football players at the FIFA U-20 and U-17 Women's World Cup 2022.

Exclusion Criteria:

* No exclusion criteria are present except refusal to provide consent for data to me used in this study.

Ages: 15 Years to 20 Years | Sex: Female
Age Groups: Child, Adult
Study Population: This research project will be performed at the FIFA U-20 Women's World Cup 2022 final tournament which is played in Alajuela and San José, Costa Rica between August 10 and August 28, 2022, and the FIFA U-17 Women's World Cup 2022 final tournament which is played in Bhubaneswar, Goa, and Navi Mumbai, India between October 11 and October 30th, 2022.
  Each tournament includes 16 national teams, and each team is allowed to select 21 players, giving at total of 336 potential participants per tournament. In total, 32 matches will be played over 19 days, with the 24 group stage matches played in the first 8 days and the 8 knock-out matches played in the last 9 days.
Sampling Method: Probability Sample
Enrollment: 672 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Time-loss injury | August 2022
  * Time-loss is defined as inability of a player to complete the current or future training session or match.
  * Injury is defined as tissue damage or other derangement of normal physical function resulting from rapid or repetitive transfer of kinetic energy.
Time-loss illness | October 2022
  * Time-loss is defined as inability of a player to complete the current or future training session or match.
  * Illness is defined as a health-related complaint or disorder experienced by an athlete, not considered as an injury.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Serner, PhD, Principal Investigator — Fédération Internationale de Football Association
Locations (1):
- Fèdèration Internationale de Football Association, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No